CLINICAL TRIAL: NCT04511650
Title: Phase 2, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Dose Escalation and Proof-of-Concept Study to Evaluate the Safety and Efficacy of Razuprotafib in Hospitalized Subjects With Coronavirus Disease 2019
Brief Title: Evaluation of the Safety and Efficacy of Razuprotafib in Hospitalized Subjects With Coronavirus Disease 2019
Acronym: RESCUE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: After completion of Step 1 Part 1, the Sponsor discontinued the study based on challenges associated with recruiting and monitoring patients in the current pandemic environment.
Sponsor: EyePoint Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: AKB-9778-CI-6001
Record Dates: First submitted 2020-08-07; First posted 2020-08-13 (Actual); Results first posted 2023-06-08 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: COVID-19; Acute Respiratory Distress Syndrome (ARDS)
Keywords: COVID-19; ARDS; Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2)
MeSH Terms: conditions — COVID-19; Respiratory Distress Syndrome | interventions — Solutions

STUDY DESIGN:
Intervention Model Description: The study was planned to include 2 parts with Part 1 comprising the dose escalation period of the study and Part 2 comprising the proof-of-concept safety and efficacy period of the study. Although The Data Review Committee (DRC) recommended to continue with the study after the completion of Part 1, Step 1, the Sponsor elected to discontinue the study due to business-related reasons.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Razuprotafib 10 mg (Experimental): Active Comparator
  Interventions: Drug: Razuprotafib Subcutaneous Solution
- Placebo (Placebo Comparator): Placebo Comparator
  Interventions: Drug: Placebo Subcutaneous Solution
- Razuprotafib 20 mg (Experimental): Active Comparator
  Interventions: Drug: Razuprotafib Subcutaneous Solution

INTERVENTIONS:
Drug: Razuprotafib Subcutaneous Solution — Up to 3 daily dose levels of Razuprotafib Subcutaneous Solution will be evaluated. Doses will be administered subcutaneously three times daily (Q8H) for 7 days.
  Other Names: Razuprotafib 10 mg and 20 mg solution
  Arms: Razuprotafib 10 mg; Razuprotafib 20 mg
Drug: Placebo Subcutaneous Solution — Matched vehicle-controlled placebo solution will be administered subcutaneously three times daily (Q8H) for 7 days
  Other Names: Placebo comparator
  Arms: Placebo

SUMMARY:
This was a Phase 2, randomized, double-blind, placebo-controlled, parallel-group, multicenter, dose escalation and proof-of-concept study to evaluate the safety and efficacy of razuprotafib, administered 3 times daily (TID) (every 8 hours [Q8H]), in hospitalized subjects with moderate to severe Coronavirus disease 2019 (COVID-19) receiving standard of care therapy.

The study was planned to include 2 parts with Part 1 comprising the dose escalation period of the study and Part 2 comprising the proof-of-concept safety and efficacy period of the study.

DETAILED DESCRIPTION:
Part 1 was to be a 2-step dose escalation that included approximately 60 subjects. Part 1, Step 1 was to include 30 subjects, and Part 1, Step 2 was to include 30 subjects. Part 1 was designed to primarily focus on safety; however, efficacy data was to be collected and analyzed as well.

Despite the Data Review Committee (DRC) recommendation to continue the study, after completion of Part 1, Step 1, the Sponsor elected to discontinue the study due to business-related reasons. Recruitment challenges and slow site startup led to delays in completing the study in a practical timeframe, and were the primary reasons to discontinue the study. No further subjects were recruited after Part 1, Step 1 completion. A full analysis of the data from Part 1, Step 1 was conducted and is presented in this report.

Part 1, Step 2 and Part 2 was not conducted.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and provide informed consent;
2. Males and non-pregnant females 18 years of age or older at the time of Screening;
3. Laboratory-confirmed active SARS-CoV-2 infection within 72 hours prior to randomization, or (if testing results cannot be obtained) by evidence of progressive disease suggestive of ongoing SARS-CoV-2 infection;
4. Females of childbearing potential must be willing to completely abstain or agree to use a highly effective method of contraception through Day 28; and have a negative urine pregnancy test during Screening;
5. Currently hospitalized, receiving standard of care therapy for COVID-19, and meets the criteria for moderate or severe COVID-19, as follows: Moderate = symptoms of moderate illness with COVID-19, which could include any symptom of mild illness or shortness of breath with exertion and with respiratory rate at 20 or greater breaths/min, Peripheral capillary oxygen saturation (SpO2) >93% on room air at sea level, or heart rate at 90 or greater beats/min; Severe = symptoms suggestive of severe systemic illness with COVID-19, which could include any symptom of moderate illness, shortness of breath at rest, or respiratory distress, and respiratory rate at 30 or greater breaths/min, heart rate at 125 or greater beats/min, or SpO2 >93% on room air at sea level or (partial pressure of oxygen:fraction of inspired oxygen (PaO2:FiO2) <300.

Exclusion Criteria:

1. Inability to initiate study drug within 12 hours after randomization;
2. Female of childbearing potential who is unable or unwilling to forego breastfeeding through Day 28;
3. Systolic blood pressure <100 mmHg;
4. In shock or requiring pressor support;
5. Respiratory failure, defined as subjects who are on mechanical ventilation; are receiving oxygen delivered by high-flow nasal cannula (heated, humidified, oxygen delivered via reinforced nasal cannula at flow rates >20 L/min with fraction of delivered oxygen of 0.5 or greater), noninvasive positive pressure ventilation, or extracorporeal membrane oxygenation (ECMO); or have a clinical diagnosis of respiratory failure (ie, clinical need for 1 of the preceding therapies, but preceding therapies not able to be administered in setting of resource limitation);
6. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >3 × the upper limit of normal (ULN);
7. Total bilirubin >2 × ULN;
8. Estimated glomerular filtration rate <30 mL/min or receiving hemodialysis or hemofiltration;
9. Moribund subject not expected to survive 24 hours in the opinion of the treating clinical team;
10. Any concurrent serious medical condition (eg, active malignancies on chemotherapy, post organ transplant, end stage congestive heart failure) or not likely to respond to treatment;
11. Decision to withhold life-sustaining treatment; Note: In the event of cardiac arrest, the decision to withhold cardiopulmonary resuscitation only does not fulfill this exclusion criterion.
12. Use of cytochrome P450 (CYP) 2 subfamily C, polypeptide 8 (2C8) substrates (eg, repaglinide, paclitaxel, or cerivastatin) or CYP3A4 substrates (eg, amlodipine, budesonide, dasabuvir, enzalutamide, imatinib, lopinavir, loperamide, saquinavir, sildenafil, midazolam, or montelukast);
13. Use of CYP2C8 inhibitors (eg, gemfibrozil, fluvoxamine, or ketoconazole);
14. Participation in another investigational study during the present study through the last visit (Day 28); or
15. Previous randomization in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2020-10-21 (Actual); Primary Completion 2021-02-26 (Actual); Study Completion 2021-02-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - University of Southern California, Los Angeles, California
  - University of California- Irvine Medical Center, Orange, California
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Snake River Research, Idaho Falls, Idaho
  - University of Minnesota, Minneapolis, Minnesota
  - University of Cincinnati, Cincinnati, Ohio
  - Rhode Island Hospital, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 31 subjects (11 in the placebo, 10 in the 10 mg Razuprotafib, and 10 in the 20 mg razuprotafib groups) were enrolled from a period October 21, 2020 to February 26, 2021.
  A total of 29 subjects (10 in the placebo, 9 in the 10 mg Razuprotafib, and 10 in the razuprotafib groups) were treated with study treatment. Two subjects (1 in each of placebo and 10 mg razuprotafib groups) were randomized and not treated.
  Therefore, a total of 29 subjects are included in the safety population.
Groups:
- Razuprotafib 10 mg: Razuprotafib 10 mg Subcutaneous Solution: Up to 3 daily dose levels of Razuprotafib Subcutaneous Solution will be evaluated. Doses will be administered subcutaneously three times daily (Q8H) for 7 days.
- Razuprotafib 20 mg: Razuprotafib 20 mg Subcutaneous Solution: Up to 3 daily dose levels of Razuprotafib Subcutaneous Solution will be evaluated. Doses will be administered subcutaneously three times daily (Q8H) for 7 days.
Period: Overall Study
Arm/Group | Razuprotafib 10 mg | Razuprotafib 20 mg | Placebo
Started | 10 | 10 | 11
Subjects Treated | 9 | 10 | 10
Subjects Randomized But Not Treated | 1 | 0 | 1
Completed | 7 | 9 | 9
Not Completed | 3 | 1 | 2
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — reason not provided | 0 | 0 | 1
Not completed — Death | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Razuprotafib 10mg; Razuprotafib 20mg: Razuprotafib Subcutaneous Solution: Up to 3 daily dose levels of Razuprotafib Subcutaneous Solution will be evaluated. Doses will be administered subcutaneously three times daily (Q8H) for 7 days.
- Total: Total of all reporting groups
Arm/Group | Razuprotafib 10mg | Razuprotafib 20mg | Placebo | Total
Number analyzed (Participants) | 10 | 10 | 11 | 31
Age, Customized [Mean (Standard Deviation); unit: years]
  Age at Informed Consent | 58.3 (11.52) | 53.4 (16.55) | 62.7 (15.81) | 58.3 (14.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 5 | 8
  Male | 9 | 8 | 6 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 0 | 7
  Not Hispanic or Latino | 5 | 7 | 11 | 23
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 3 | 0 | 3 | 6
  White | 4 | 7 | 8 | 19
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 0 | 3
Coronavirus disease (COVID-19) severity, n (%) [Count of Participants; unit: Participants] — Moderate COVID-19: (1) Symptoms which could include shortness of breath with exertion, fever, dry cough, headache, body aches, chills, loss of taste or smell; and (2) respiratory rate of >= 20 breaths/min, oxygen saturation >93% on room air at sea level, or heart rate >=90 bts/min.
  Severe COVID-19: (1) symptoms which could include shortness of breath at rest or respiratory distress; and (2) Respiratory rate >=30 breaths/min, heart rate >= 125 bts/min, or oxygen saturation <=93% on room air at sea level or partial oxygen:fraction of inspired oxygen <300
  Participants
    Moderate | 3 | 2 | 3 | 8
    Severe | 7 | 8 | 8 | 23
National Institutes of Allergy and Infectious Diseases [Count of Participants; unit: Participants] — The National Institute of Allergy and Infectious Disease (NIAID) 8-Point Scale is an 8-point ordinal scale. The NIAID score was a measured the subjects clinical status at baseline at each study visit. The NIAID assessment at baseline was summarized by the number and percent of subjects for each of the 8 categories was summarized by treatment group and overall.
  Participants
    Category 1 = Death | 0 | 0 | 0 | 0
    Category 2 = Hospitalized on mechanical ventilation | 0 | 0 | 0 | 0
    Category 3 = Hospitalized, on noninvasive ventilation or high-flow oxygen devices | 4 | 5 | 4 | 13
    Category 4= Hospitalized, requiring supplemental oxygen | 5 | 5 | 6 | 16
    Category 5= Hospitalized, not requiring supplemental oxygen - requiring ongoing COVID-19 care | 1 | 0 | 1 | 2
    Category 6= Hospitalized, not requiring supplemental oxygen - no longer requires medical care | 0 | 0 | 0 | 0
    Category 7=Not hospitalized, limitation on activities or requiring home oxygen | 0 | 0 | 0 | 0
    Category 8= Not hospitalized, no limitations on activities | 0 | 0 | 0 | 0
Screening Peripheral Oxygen Saturation (Pa02)/Fraction of Inspired Oxygen (FiO2) ratio [Mean (Standard Deviation); unit: ratio] — Population: n= the number of participants included in the ratio mean (SD) calculation as shown in Table 3 of the demographics and baseline characteristics table for the ITT population.
  One subject in each of the Razuprotafib 10mg and placebo group were randomized and not treated; therefore, these two subjects are not included in the analyses.
  ratio
    number analyzed (Participants) | 9 | 9 | 10 | 28
    (all) | 194.97 (131.546) | 146.15 (80.602) | 212.40 (132.210) | 186.71 (118.212)
Pre-hospitalization oxygen requirement, n (%) [Count of Participants; unit: Participants]
  None | 7 | 10 | 10 | 27
  Low-flow nasal cannula | 2 | 0 | 1 | 3
  CPAP mask (for non-respiratory failure reasons) | 1 | 0 | 0 | 1
Concomitant medications to treat COVID-19 at baseline, n (%) [Count of Participants; unit: Participants] — participants may have been receiving more than one concomitant medication listed and therefore, the total N will not add up to the n.
  Participants
    Remdesivir | 3 | 6 | 8 | 17
    Systemic steroids | 8 | 10 | 10 | 28
    Other | 6 | 8 | 4 | 18
    None | 1 | 0 | 1 | 2
Comorbid conditions, n (%) [Count of Participants; unit: Participants]
  Diabetes | 3 | 4 | 6 | 13
  Obesity | 4 | 4 | 2 | 10
  Hypertension | 8 | 6 | 5 | 19
  Heart Failure | 1 | 0 | 0 | 1
  Chronic Kidney Disease | 1 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number and Percent of Subjects Who Were Alive and Free of Respiratory Failure Prior to Day 7 and Day 28
Description: All results were summarized descriptively by treatment arm and expressed as proportions, along with corresponding 95%CI of the difference between response rates, and p-values using Cochran-Mantel-Haenszel (CMH). The 95% CI will be constructed using the normal approximation method. Respiratory failure was defined as subjects who were on invasive mechanical ventilation; received oxygen delivered by high-flow nasal cannula (heated, humidified, oxygen delivered via reinforced nasal cannula at flow rates >20L/min with fraction of delivered oxygen ≥0.5) noninvasive positive pressure ventilation or extracorporeal membrane oxygenation; or had a clinical diagnosis of respiratory failure (ie, clinical need for 1 of the preceding therapies, but preceding therapies not able to be administered in setting of resource limitation).Subjects who died prior to the study timepoint (Day 7 or Day 28) were imputed based on the worst outcome.
Time Frame: Baseline up to Day 7 and Day 28
Population: The Full Analysis (FA) Population included subjects who received at least 1 dose of study drug and had at least 1 post-dose efficacy evaluation. The FA Population was a subset of the ITT Population which was defined as all subjects randomized. Note: The overall number of participants analyzed represents the total number of participants in each treatment group for the FA Population. Count of participants who were alive and free of respiratory failure on Days 7 and 28 were included in analyses.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Placebo for razuprotafib was sterile normal saline
- Pooled Razuprotafib: Razuprotafib 10 and 20 mg pooled
Arm/Group | Placebo | Razuprotafib 10 mg | Razuprotafib 20 mg | Pooled Razuprotafib
Number analyzed (Participants) | 10 | 9 | 10 | 19
Participants
  Number and Percent of Subjects who were Alive and Free of Respiratory Failure Prior to Day 7 | 8 | 5 | 6 | 11
  Number and Percent of Subjects who were Alive and Free of Respiratory Failure Prior to Day 28: number analyzed (Participants) | 10 | 8 | 10 | 18
  Number and Percent of Subjects who were Alive and Free of Respiratory Failure Prior to Day 28 | 9 | 6 | 7 | 13

2. Secondary Outcome: Summary of The Mean Change From Baseline in D-Dimer at Day 7 and 28
Description: Mean Change from baseline in systemic biomarkers of vascular leakage and inflammation (ie, D-Dimer) at Day 7 and 28 in the Full Analysis Set
Time Frame: at Day 7 and 28
Population: Full Analysis (FA) Population: The FA Population was a subset of the ITT Population and included subjects who received at least 1 dose of study drug and had at least 1 post-dose efficacy evaluation. Note: The overall number of participants analyzed represents the total number of participants in each treatment group for the FA Population. The summaries of the mean change from baseline analyses included those participants who had post-baseline D-Dimer values available on Days 7 and 28.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo | Razuprotafib 10 mg | Razuprotafib 20 mg
Number analyzed (Participants) | 10 | 9 | 10
ng/mL
  Baseline: number analyzed (Participants) | 10 | 8 | 10
  Baseline | 466.9 (243.85) | 1750.9 (2137.46) | 823.2 (787.39)
  Mean Change from Baseline at Day 7 | -144.5 (133.63) | 8913.4 (16869.43) | 2239.0 (5485.79)
  Mean change from baseline at Day 28: number analyzed (Participants) | 0 | 0 | 2
  Mean change from baseline at Day 28 |  |  | 2121.0 (1566.95)

3. Secondary Outcome: Summary of Change From Baseline in C-Reactive Protein (CRP) at Day 7 and 28
Description: Change from baseline in systemic biomarkers of vascular leakage and inflammation (ie, CRP ) at Day 7 and 28 in the Full Analysis Set
Time Frame: at Day 7 and 28
Population: Full Analysis (FA) Population: The FA Population was a subset of the ITT Population and included subjects who received at least 1 dose of study drug and had at least 1 post-dose efficacy evaluation. Note: The overall number of participants analyzed represents the total number of participants in each treatment group for the FA Population. The summaries of the mean change from baseline analyses included those participants who had post-baseline CRP values available on Days 7 and 28.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Razuprotafib 10 mg | Razuprotafib 20 mg
Number analyzed (Participants) | 10 | 9 | 10
mg/dL
  Baseline: number analyzed (Participants) | 9 | 8 | 9
  Baseline | 17.44 (27.17) | 25.67 (50.64) | 23.01 (45.95)
  Mean Change from Baseline at Day 7: number analyzed (Participants) | 8 | 5 | 8
  Mean Change from Baseline at Day 7 | -13.17 (21.80) | -29.55 (60.99) | -22.64 (47.95)
  Mean change from baseline at Day 28: number analyzed (Participants) | 0 | 0 | 2
  Mean change from baseline at Day 28 |  |  | -4.26 (3.87)

4. Secondary Outcome: Number of Participants Who Improve by at Least 2 Categories on the NIAID 8-point Ordinal Scale From Baseline to Day 7 and Baseline to Day 28
Description: Analysis of the proportion of participants who improve by >=2 categories on the NIAID 8-point scale from baseline to Day 7. % = 100 x n/N', where N' = number of participants with a non-missing values at baseline and the specified post-baseline visit. Baseline is defined as the last measurement prior to the first dose of study drug.
Time Frame: from baseline to Day 7 and baseline to Day 28
Population: Full Analysis (FA) Population: The FA Population was a subset of the ITT Population and included participants who received at least 1 dose of study drug and had at least 1 post-dose efficacy evaluation. Note: The overall number of participants analyzed represents the total number of participants in each treatment group for the FA Population. The count of participants who had NIAID 8-point scale results at the Day 7 and Day 28 timepoints were included in the analyses.
Measure: Count of Participants; unit: Participants
Groups:
- Pooled Razuprotafib: Subjects treated with Razuprotafib 10 and 20 mg.
Arm/Group | Placebo | Razuprotafib 10 mg | Razuprotafib 20 mg | Pooled Razuprotafib
Number analyzed (Participants) | 10 | 9 | 10 | 19
Participants
  Participants who improved by >=2 categories from Baseline to Day 7: number analyzed (Participants) | 8 | 7 | 8 | 15
  Participants who improved by >=2 categories from Baseline to Day 7 | 5 | 2 | 2 | 4
  Subjects who improved by >=2 categories from Baseline to Day 28: number analyzed (Participants) | 10 | 8 | 10 | 18
  Subjects who improved by >=2 categories from Baseline to Day 28 | 9 | 6 | 7 | 13

5. Secondary Outcome: Number of Participants Who Were Discharged and Free of Respiratory Failure Prior to Day 7 and Day 28
Description: The number of participants who were discharged and free of respiratory failure at Day 7 and Day 28 were summarized by treatment arm and pooled razuprotafib (10 and 20 mg) group.
Time Frame: Day 7 and Day 28
Population: Full Analysis (FA) Population: The FA Population was a subset of the ITT Population and included participants who received at least 1 dose of study drug and had at least 1 post-dose efficacy evaluation. Note: The overall number of participants analyzed represents the total number of participants in each treatment group for the FA Population. The count of participants who were discharged and free of respiratory failure at the Day 7 and Day 28 timepoints.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Placebo is sterile normal saline
- Pooled Razuprotafib: pooled 10 and 20 mg Razuprotafib groups
Arm/Group | Placebo | Razuprotafib 10 mg | Razuprotafib 20 mg | Pooled Razuprotafib
Number analyzed (Participants) | 10 | 9 | 10 | 19
Participants
  Prior to Day 7 | 7 | 3 | 4 | 7
  Prior to Day 28: number analyzed (Participants) | 9 | 7 | 9 | 16
  Prior to Day 28 | 9 | 6 | 7 | 13

6. Secondary Outcome: Number of Participants Alive and Not Requiring Invasive Mechanical Ventilation at Any Time
Description: Analysis of Number of Participants Alive and Not Requiring Invasive Mechanical Ventilation at Any Time Through Day 28 in the Full Analysis Set
Time Frame: Baseline up to Day 28
Population: Full Analysis (FA) Population: The FA Population was a subset of the ITT Population and included participants who received at least 1 dose of study drug and had at least 1 post-dose efficacy evaluation. Note: The overall number of participants analyzed represents the total number of participants in each treatment group for the FA Population. The count of participants who had post-baseline data and were alive and not requiring mechanical ventilation were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Razuprotafib 10 mg | Razuprotafib 20 mg | Pooled Razuprotafib
Number analyzed (Participants) | 10 | 8 | 10 | 18
Participants | 9 | 6 | 8 | 14
Statistical Analysis 1: Comparison: Placebo vs Pooled Razuprotafib; Pooled Razuprotafib comparison to Placebo. All results are summarized descriptively by treatment arm and expressed as proportions, along with corresponding 95% confidence intervals (CIs) of the difference between response rates, and p-values; Test type: Superiority; p = 0.4795, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test stratified by disease severity

7. Secondary Outcome: Time to Reach Grade 6, 7, or 8 on the NIAID 8-Point Ordinal Scale
Description: The clinical status of the participants was assessed within 1 hr prior to each dose of study drug, using the NIAID 8-point ordinal scale until Day 28. After the treatment period, clinical status will be assessed once daily until Day 18, unless discharged. If the subject is discharged alive prior to Day 28, clinical status was assessed at the post-treatment observation period telephone visits only. Grade 6=hospitalized, not requiring oxygen and no longer requires ongoing medical care; Grade 7 = not hospitalized, limitation on activities and/or requiring home oxygen; and Grade 8 = not hospitalized, no limitations on activities.
Time Frame: From Screening through the end of the study (up to 28 days)
Population: Intent-to-Treat (ITT) Population: The ITT Population was defined as all subjects randomized. Participants in this population were analyzed according to the treatment group to which they were assigned at randomization. Note: The overall number of participants analyzed represents the total number of participants in each treatment group for the ITT Population. The number of participants included in the analyses had post-baseline data through the end of the study.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo | Razuprotafib 10 mg | Razuprotafib 20 mg | Pooled Razuprotafib
Number analyzed (Participants) | 9 | 7 | 7 | 14
days | 9.8 (5.87) | 11.7 (7.87) | 11.7 (5.47) | 11.7 (6.51)

8. Secondary Outcome: Change in PaO2:FiO2 Ratio From Baseline to Day 7 and Baseline to Day 28
Description: Analysis of the change in PaO2:FiO2 ratio from baseline to Day 7 (or discharge) and baseline to Day 28 (or discharge) in the intent-to-treat population. Baseline was defined as the last measurement prior to the first dose of study drug. Baseline PaO2;FiO2 ratio value was not provided for the pooled Razuprotafib group.
Time Frame: Baseline up to Day 7 and Day 28
Population: Intent-to-Treat (ITT) Population: The ITT Population was defined as all subjects randomized. Participants in this population were analyzed according to the treatment group to which they were assigned at randomization. Note: The overall number of participants analyzed represents the total number of participants in each treatment group for the ITT Population. The summaries of the mean changes from baseline included only those participants with available data.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Placebo | Razuprotafib 10 mg | Razuprotafib 20 mg | Pooled Razuprotafib
Number analyzed (Participants) | 11 | 10 | 10 | 20
ratio
  Baseline: number analyzed (Participants) | 11 | 10 | 9 | 0
  Baseline | 212.40 (132.210) | 194.97 (131.546) | 146.15 (80.602) |
  Day 7: number analyzed (Participants) | 5 | 5 | 6 | 11
  Day 7 | 27.44 (55.259) | 18.81 (82.833) | 48.34 (81.008) | 34.92 (79.142)
  Day 28: number analyzed (Participants) | 4 | 2 | 4 | 6
  Day 28 | 140.95 (76.887) | 96.21 (155.077) | 117.01 (87.030) | 110.08 (97.312)

9. Secondary Outcome: Length of Hospitalization and Not Requiring Invasive Mechanical Ventilation From Baseline to Day 7 and Day 28 (or Death)
Description: Analysis of length of hospitalization and not requiring invasive mechanical ventilation from baseline to Day 7 and Day 28 in the intent-to-treat population. Note: The overall number of participants analyzed represents the total number of participants in each treatment group for the ITT Population. The summaries of the mean number of days from baseline included only those participants with available data. Baseline was defined as the last measurement prior to the first dose of study drug. Baseline values were not provided.The length of hospitalization was to include all days that the participant was admitted to the hospital. For participants who were discharged and readmitted to the hospital, the length of hospitalization was to include the days after readmission. Hospitalization days were counted in 24-hour periods; any partial days were counted as a whole day.
Time Frame: Baseline up to Day 7 and Day 28
Population: Intent-to-Treat (ITT) Population: The ITT Population was defined as all subjects randomized. Participants in this population were analyzed according to the treatment group to which they were assigned at randomization. Note: The overall number of participants analyzed represents the total number of participants in each treatment group for the ITT Population. Those participants who had post-baseline values on Day 7 and 28 were included in the analyses.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Placebo | Razuprotafib 10 mg | Razuprotafib 20 mg | Pooled Razuprotafib
Number analyzed (Participants) | 11 | 10 | 10 | 20
Days
  Day 7: number analyzed (Participants) | 10 | 9 | 10 | 19
  Day 7 | 5.0 (1.70) | 5.8 (2.17) | 6.2 (1.14) | 6.0 (1.67)
  Day 28: number analyzed (Participants) | 10 | 8 | 10 | 18
  Day 28 | 7.2 (4.69) | 9.9 (6.64) | 12.7 (8.31) | 11.4 (7.54)

10. Secondary Outcome: Length of Hospitalization From Baseline to Day 7 and Day 28 (or Death)
Description: Analysis of length of hospitalization from baseline to day 7 and day 28 (or death) in the intent-to-treat population. Baseline was defined as the last measurement prior to the first dose of study drug. Baseline values were not provided. The length of hospitalization was to include all days that the participant was admitted to the hospital. For participants who were discharged and readmitted to the hospital, the length of hospitalization was to include the days after readmission. Hospitalization days were counted in 24-hour periods; any partial days were counted as a whole day.
Time Frame: From Baseline to Day 7 or Day 28 (or Death)
Population: Intent-to-Treat (ITT) Population: The ITT Population was defined as all subjects randomized. Participants in this population were analyzed according to the treatment group to which they were assigned at randomization. Note: The overall number of participants analyzed represents the total number of participants in each treatment group for the ITT Population. Participants who had post-baseline data on Days 7 and 28 (or death) were included in the analyses.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Placebo | Razuprotafib 10 mg | Razuprotafib 20 mg | Pooled Razuprotafib
Number analyzed (Participants) | 11 | 10 | 10 | 20
Days
  Day 7: number analyzed (Participants) | 10 | 9 | 10 | 19
  Day 7 | 5.0 (1.70) | 5.8 (2.17) | 6.2 (1.14) | 6.0 (1.67)
  Day 28: number analyzed (Participants) | 10 | 8 | 10 | 18
  Day 28 | 7.2 (4.69) | 14.1 (9.69) | 14.6 (9.47) | 14.4 (9.28)

11. Secondary Outcome: Number of Participants Who Worsen by Greater Than or Equal to 2 Categories on The NIAID 8-point Ordinal Scale From Baseline to Day 7 and Day 28
Description: Analysis of number of participants who worsen by >= 2 categories on the NIAID 8-point ordinal scale from baseline to Day 7 in the Full Analysis Population. % = 100 x n/N', where N' = number of participants with non-missing values at baseline and the specified post-baseline visit. Participants who died prior to the Day 7 or Day 28 were imputed as 1.
Time Frame: From baseline to Day 7 and Day 28
Population: Full Analysis (FA) Population: The FA Population was a subset of the ITT Population and included participants who received at least 1 dose of study drug and had at least 1 post-dose efficacy evaluation. Note: The overall number of participants analyzed represents the total number of participants in each treatment group for the FA Population. Those participants who had post-baseline data on Days 7 and 28 were included in the analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Razuprotafib 10 mg | Razuprotafib 20 mg | Pooled Razuprotafib
Number analyzed (Participants) | 10 | 9 | 10 | 19
Participants
  Participants who worsened by >= 2 categories from baseline to Day 7: number analyzed (Participants) | 8 | 7 | 8 | 19
  Participants who worsened by >= 2 categories from baseline to Day 7 | 0 | 0 | 0 | 0
  Participants who worsened by >= 2 categories from baseline to Day 28: number analyzed (Participants) | 10 | 8 | 10 | 18
  Participants who worsened by >= 2 categories from baseline to Day 28 | 1 | 1 | 1 | 2

12. Secondary Outcome: Number of Participants in Each Category of the NIAID 8-point Ordinal Scale at Day 7 and Day 28
Description: Summary of number and percent of subjects in each category (ie, categories 1 to 8) of the NIAID 8-Point Ordinal Scale at baseline, Day 7 and Day 28. The NIAID 8-point ordinal scale includes the following grades:
  1. Death;
  2. Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO);
  3. Hospitalized, on noninvasive ventilation or high-flow oxygen devices;
  4. Hospitalized, requiring supplemental oxygen;
  5. Hospitalized, not requiring supplementation oxygen - requiring ongoing medical care (COVID-19 related or otherwise);
  6. Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care;
  7. Not hospitalized, limitation on activities and/or requiring home oxygen; and
  8. Not hospitalized, no limitations on activities.
Time Frame: Baseline, Day 7, and Day 28
Population: Intent-to-Treat (ITT) Population: The ITT Population was defined as all subjects randomized. Subjects in this population were analyzed according to the treatment group to which they were randomized. Note: The overall number of participants analyzed represents the total number of participants in each treatment group for the ITT Population. Those participants who had Baseline and post-baseline data on Days 7 and 28 were included in the analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Razuprotafib 10 mg | Razuprotafib 20 mg | Pooled Razuprotafib
Number analyzed (Participants) | 11 | 10 | 10 | 20
Participants
  Baseline: number analyzed (Participants) | 10 | 9 | 10 | 19
  Baseline: 1 | 0 | 0 | 0 | 0
  Baseline: 2 | 0 | 0 | 0 | 0
  Baseline: 3 | 4 | 4 | 6 | 10
  Baseline: 4 | 6 | 4 | 4 | 8
  Baseline: 5 | 0 | 1 | 0 | 1
  Baseline: 6 | 0 | 0 | 0 | 0
  Baseline: 7 | 0 | 0 | 0 | 0
  Baseline: 8 | 0 | 0 | 0 | 0
  Day 7: number analyzed (Participants) | 8 | 7 | 8 | 15
  Day 7: 1 | 0 | 0 | 0 | 0
  Day 7: 2 | 0 | 0 | 0 | 0
  Day 7: 3 | 2 | 4 | 4 | 8
  Day 7: 4 | 1 | 1 | 2 | 3
  Day 7: 5 | 0 | 0 | 0 | 0
  Day 7: 6 | 0 | 0 | 0 | 0
  Day 7: 7 | 4 | 1 | 1 | 2
  Day 7: 8 | 1 | 1 | 1 | 2
  Day 28: number analyzed (Participants) | 9 | 7 | 9 | 16
  Day 28: 1 | 0 | 0 | 0 | 0
  Day 28: 2 | 0 | 1 | 1 | 2
  Day 28: 3 | 0 | 0 | 1 | 1
  Day 28: 4 | 0 | 0 | 0 | 0
  Day 28: 5 | 0 | 0 | 0 | 0
  Day 28: 6 | 0 | 0 | 0 | 0
  Day 28: 7 | 5 | 3 | 5 | 8
  Day 28: 8 | 4 | 3 | 2 | 5

13. Secondary Outcome: The Number and Percent of Participants Who Experienced All-Cause Mortality at Day 7 and Day 28
Description: Analysis of the Number and Percent of Participants who Experienced All-Cause Mortality at Day 7 and Day 28 in the Full Analysis Set
Time Frame: Baseline up to Day 7 and Day 28
Population: Full Analysis (FA) Population: The FA Population was a subset of the ITT Population and included subjects who received at least 1 dose of study drug and had at least 1 post-dose efficacy evaluation. Note: The overall number of participants analyzed represents the total number of participants in each treatment group for the FA Population. The participants who had post-baseline data on Days 7 and 28 were included in the all-cause mortality analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Razuprotafib 10 mg | Razuprotafib 20 mg | Pooled Razuprotafib
Number analyzed (Participants) | 10 | 9 | 10 | 19
Participants
  All-Cause Mortality at Day 7 | 0 | 0 | 0 | 0
  All-Cause Mortality at Day 28: number analyzed (Participants) | 10 | 8 | 10 | 18
  All-Cause Mortality at Day 28 | 1 | 1 | 1 | 2

14. Secondary Outcome: Number of Participants Who Improve by Greater or Equal to 2 Categories on the NIAID 8-point Ordinal Scale From Baseline to Day 7 and Day 28
Description: Analysis of number of participants who improve by >= 2 categories on the NIAID 8-point scale from baseline to Day 7 and Day 28 in the full analysis set.% = 100 x n/N', where N' = number of participants with non-missing values at baseline and the specified post-baseline visit. Participants who died prior to the Day 7 or Day 28 were imputed as 1.
Time Frame: Baseline to Day 7 and Day 28
Population: Full Analysis (FA) Population: The FA Population was a subset of the ITT Population and included participants who received at least 1 dose of study drug and had at least 1 post-dose efficacy evaluation. Note: The overall number of participants analyzed represents the total number of participants in each treatment group for the FA Population. Those participants who had post-baseline data on Day 7 and 28 were included in analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Razuprotafib 10 mg | Razuprotafib 20 mg | Pooled Razuprotafib
Number analyzed (Participants) | 10 | 9 | 10 | 19
Participants
  Participants who improve by >=2 categories on Day 7: number analyzed (Participants) | 8 | 7 | 8 | 15
  Participants who improve by >=2 categories on Day 7 | 5 | 2 | 2 | 4
  Participants who improve by >=2 categories on Day 28: number analyzed (Participants) | 10 | 8 | 10 | 18
  Participants who improve by >=2 categories on Day 28 | 9 | 6 | 7 | 13

15. Secondary Outcome: Time to Return to Prehospitalization Oxygen Requirement
Description: Summary of Time to Return to Prehospitalization Oxygen Requirement in the Intent-to-Treat Population
Time Frame: up to 28 days
Population: Intent-to-Treat (ITT) Population: The ITT Population was defined as all participants randomized. Participants in this population were analyzed according to the treatment group to which they were assigned at randomization.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Placebo | Razuprotafib 10 mg | Razuprotafib 20 mg | Pooled Razuprotafib
Number analyzed (Participants) | 7 | 7 | 3 | 10
Days | 5.1 (5.05) | 6.4 (7.83) | 9.7 (9.87) | 7.4 (8.06)

16. Other Pre Specified Outcome: Summary of Razuprotafib Plasma Concentration
Description: A summary of plasma razuprotafib concentrations for samples collected on Day 1 and 6 in the pharmacokinetic population. All results were summarized descriptively by treatment group.
Time Frame: razuprotafib plasma concentrations 30 and 90 minutes post-dose on Days 1 and 6
Population: Pharmacokinetic (PK) Population: The PK Population was defined as all randomized subjects who received at least 1 dose of study drug and had least 1 PK sample with plasma concentration.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo | Razuprotafib 10 mg | Razuprotafib 20 mg
Number analyzed (Participants) | 0 | 9 | 10
ng/mL
  Razuprotafib Plasma Concentration 30 minutes post-dose on Day 1: number analyzed (Participants) | 0 | 9 | 9
  Razuprotafib Plasma Concentration 30 minutes post-dose on Day 1 |  | 87.88 (33.24) | 194.73 (67.20)
  Razuprotafib plasma concentration 90 minutes post-dose on Day 1 |  | 64.68 (21.29) | 124.57 (33.88)
  Razuprotafib Plasma Concentration 30 minutes post-dose on Day 6: number analyzed (Participants) | 0 | 6 | 4
  Razuprotafib Plasma Concentration 30 minutes post-dose on Day 6 |  | 64.98 (41.03) | 105.82 (71.99)
  Razuprotafib Plasma Concentration 90 minutes post-dose on Day 6: number analyzed (Participants) | 0 | 6 | 4
  Razuprotafib Plasma Concentration 90 minutes post-dose on Day 6 |  | 41.04 (25.65) | 78.48 (56.13)

ADVERSE EVENTS:
Time Frame: Adverse events will be monitored at the time of screening until Day 28. Serious Adverse Events (SAEs) will be reported 30 days after the last dose of study treatment.
Arm/Group | Placebo | Razuprotafib 10 mg | Razuprotafib 20 mg
All-Cause Mortality (participants affected / at risk) | 1/10 | 1/9 | 1/10
Serious Adverse Events (participants affected / at risk) | 2/10 | 2/9 | 5/10
Other Adverse Events (participants affected / at risk) | 6/10 | 7/9 | 8/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=10) | Razuprotafib 10 mg (N=9) | Razuprotafib 20 mg (N=10)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 2 (2)
COVID-19 viral pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bacterial pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
septic shock (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
post-procedural hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Transient hypotension (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=10) | Razuprotafib 10 mg (N=9) | Razuprotafib 20 mg (N=10)
hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 2 (2)
hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
hypoproteinaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 2 (2)
Fibrin D-dimer increased (Investigations) | 0 (0) | 1 (1) | 2 (2)
White blood cell count (Investigations) | 0 (0) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 5 (5)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 3 (3) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Septic Shock (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Barotrauma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Metabolic alkalosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Blood bicarbonate increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Shock (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Neutrophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Thromobcytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Fungaemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Ischaemic hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Acquired phimosis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Product acquired from Aerpio with limited transfer of documents. Site Clinical Trial Agreements (CTAs) not provided.

DOCUMENTS (2):
  • Study Protocol (2020-12-10): https://cdn.clinicaltrials.gov/large-docs/50/NCT04511650/Prot_001.pdf
  • Statistical Analysis Plan (2021-02-16): https://cdn.clinicaltrials.gov/large-docs/50/NCT04511650/SAP_002.pdf